CLINICAL TRIAL: NCT06161649
Title: To Investigate Whether a Continuous Intelligent and Automated Mobile Education System Can Improve Knowledge, Self-care, Emotional Stress, Self-efficacy and Quality of Life in Patients With Heart Failure
Brief Title: Mobile Education System to Improve Disease Knowledge, Self-efficacy and Quality of Life in Patients With Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, MIN-HUI LIU, Heart Failure Center, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202201890B0
Record Dates: First submitted 2023-11-21; First posted 2023-12-08 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Heart failure; automation; smart mobile education system; disease knowledge; self-care; emotional stress; self-efficacy; quality of life
MeSH Terms: conditions — Heart Failure; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional outpatient care group (No Intervention): After confirming that the diagnosis of heart failure is met, the patient will receive 10-15 minutes of disease care education from a nurse when the patient receives the case. At the same time, the patient will receive a personal disease self-care education manual, and will get the contact number of the case manager in case the patients encounter emergencies or disease care needs at home (the patient can call for consultation on home care for diseases if the patient want).
- automated mobile education system group (Experimental): Intervention group (accepting the operation process of automated intelligent education software system):
  1. Execute registration and qualification review
  2. Automated smart education interaction
  At the same time, the patient will receive a personal disease self-care education manual, and will get the contact number of the case manager in case the patients encounter emergencies or disease care needs at home (the patient can call for consultation on home care for diseases if the patient want).
  Interventions: Behavioral: accepting the operation process of automated intelligent education software system

INTERVENTIONS:
Behavioral: accepting the operation process of automated intelligent education software system — 1. Execute registration and qualification review
  2. Automated smart education interaction
  Arms: automated mobile education system group

SUMMARY:
Heart failure (HF) is an incurable and complex disease syndrome with sophisticated disease trajectories. The guideline for HF management suggests that treatment should include adequate education to help patients have better self-management ability, and improve their quality of life and prognosis. However, how to provide massive amount of HF patients a continuous, complete and individualized disease care education from hospitalization, post-discharge, to home for months is a difficult problem. This study plans to develop an automated and intelligent education system for HF on the mobile device "Line" platform. Through this platform, we hope to make the HF education continuous for 3 months from hospital to post-discharge period. We hypothesize that (1) this intervention can improve knowledge, self-care, emotional stress, self-efficacy, quality of life and disease outcomes in patients of HF; (2) the system developed in this study can reduce the hours of nursing work while improve the quality of education and become the best clinical auxiliary education tool.

DETAILED DESCRIPTION:
Study background

Heart failure is a complex disease syndrome, and patients often suffer from multiple chronic diseases. Faced with the problem of disease symptoms, if patients do not have sufficient care knowledge, patients often mistakenly think that it is related to aging, and may even delay medical treatment, resulting in the need for hospitalization when it worsens. Emergency treatment may even deal with respiratory failure in severe cases. Such repeated hospitalizations will affect the quality of life and lead to poor disease prognosis for patients. Heart failure treatment guidelines have recommended that in addition to the use of standard drugs for disease treatment, systematic and structured disease education should be provided continuously during hospitalization and after discharge to help patients effectively implement disease self-management and improve the quality of disease care, quality of life and life satisfaction. Interventional studies and comprehensive literature review data have also confirmed that disease education provided by nursing staff can significantly improve the knowledge, behavior, self-efficacy, quality of life, and reduce re-hospitalization of heart failure patients. Due to the high fluctuations in the course of heart failure and the interlocking influence of multiple comorbidities, disease care information should be provided not only during hospitalization, but also during the period of discharge and at home after the acute phase. Facing complex and ever-changing disease troubles often lead to overwhelming anxiety and negative emotional stress. For heart failure patients, it is necessary to provide individualized and continuous disease care information from hospitalization, discharge to home during the chronic stage of the disease. Educational navigation helps patients have good self-efficacy to perform self-disease management at home, and then learn to coexist with the disease and obtain a better quality of life with the disease.

In recent years, during the epidemic of Coronavirus disease 2019 (COVID-19), in order to prevent the spread of the virus, disease prevention and control organizations have recommended care and management strategies for chronic diseases through remote and other mobile health care Internet platforms. Care services should be provided to maintain the continuity of nursing education in the case of zero contact. In a survey study, it was found that information sharing through social networks during the epidemic was positively helpful for patients' self-care. It can be seen that it is acceptable to use portable mobile phones for educational interaction on heart failure. Unfortunately, most of the current applications still monitor patients' physiological parameters such as blood pressure, pulse, weight, heart rhythm and other data. Mobile devices are mainly used to predict disease risk, and the provision of care information mainly uses SMS notifications to remind return visits, or simple data responses based on the results of physiological parameters. However, these require long-term measurement data to generate feedback. Since learning is a kind of interpersonal interaction, when providing disease information, if text is simply sent through text messages, patients with insufficient knowledge and literacy may not be able to identify the key points that really need to be learned. In addition, it is fixed and not personalized. The education system cannot produce substantial effects.

In the ever-changing medical environment of the epidemic, how to enable heart failure patients to continue to receive complete disease care education from hospitalization, discharge to home is a difficult problem. Because investigators have spent two years in the past working to develop an APP software platform. This platform has an automated import system, a combination of personalized educational video software, video-specific examination questions, and learning evaluation. It measures the function of the mechanism, but it still lacks intelligent performance. In addition, our heart failure center has 15 years of clinical care resources and has completed hundreds of educational videos and a tracking database of long-term patient phone interviews. Investigators hope to use cluster analysis to classify the original data. In order to explore the needs of patients at different times and achieve intelligent docking of needs and educational videos, investigators plan to develop an automated and intelligent educational assistance system for heart failure on the mobile device "Line" platform, hoping to use the assistance system in mobile devices. The intervention continues to extend heart failure disease education from the hospital to the home follow-up period, so that patients can have a sufficient disease learning process, acquire effective self-care abilities, and thereby improve their quality of life. It is also hoped that the system developed through this research can help nursing staff meet the different care needs of patients in different disease stages despite busy clinical work. Make education personal and continuous, and reduce the number of nursing work hours while still maintaining educational quality, becoming the best clinical auxiliary tool that can be replicated in education on various diseases.

The main themes of the study

1. Exploring the disease care information that heart failure patients need at different disease stages
2. Establish a continuous automated intelligent mobile education system for heart failure.
3. Participate and explore the effect of the use of continuous automated intelligent mobile education system on disease knowledge and self-care behavior of heart failure patients.
4. To explore the impact of the use of continuous automated intelligent mobile education system on anxiety and depression in patients with heart failure.
5. To explore the effectiveness of the use of continuous automated intelligent mobile education system on the self-efficacy of heart failure patients.
6. To explore the effectiveness of the use of continuous automated intelligent mobile education system on the quality of life of patients with heart failure.
7. To explore the effect of the use of continuous automated intelligent mobile education system on the six-month to one-year disease prognosis of heart failure patients.

Study Methods

According to the purpose of the research, this research plan uses a randomized controlled intervention research design method to implement and complete the research plan over a three-year period. The following is a description of the progress of the research plan in each year:

Research design Research plan This study adopts a randomized two-group pre-test and post-test experimental design to compare the effectiveness of using an automated intelligent educational software system on the self-efficacy and quality of life of patients with heart failure.

Research objects and places The first stage of this research is to complete the continuous automated intelligent mobile education system (first year). The research subjects in the second and third years of this study are selected through purposive sampling, and the subjects are patients diagnosed with heart failure in a regional teaching hospital or outpatient clinic in the north Taiwan. The conditions for inclusion and exclusion of research subjects are described in another section.

Number of samples in the second to third years In this study, participants are divided into intervention groups and control groups, and each receives five questionnaires. The estimated sample number is set with an α value of .05 and a power of .8. It is estimated that the intervention group and the control group will receive 57 cases each, totaling 114 people. It is considered that there will be a 20% attrition rate during the follow-up intervention period. Thus, the estimated sample size is 138 people.

Study tools

1. First year:

   The reliability and validity evaluation method of the educational videos in the system adopts the "Education System" developed by the Agency for Healthcare Research and Quality (AHRQ). The Patient Education Materials Assessment Tool (PEMAT) evaluates the understandability and feasibility of educational videos. This tool has two aspects, namely understandability and feasibility.
2. Two to three years:

The second phase of this study is mainly to test the effectiveness of the continuous automated intelligent mobile education system intervention program on the disease knowledge, emotional stress, self-efficacy and quality of life of heart failure patients. Structured questionnaires are adopted, including a total of six questionnaires, namely basic personal information questionnaire, heart failure knowledge scale, heart failure self-care scale, hospital anxiety and depression scale, self-efficacy scale, and quality of life scale and service satisfaction scale, as listed up below.

Intervention measures (second to third years) Introduction to the continuous automated intelligent education system: This system is developed by Liu Min Hui and Professor Wang Chao-Hung from Keelung Chang Gung Memorial Heart Failure Center.

The description of the confidentiality methods, information security measures, and database storage and management measures for network information security subjects is as follows:

1. Confidentiality of Subject Information
2. Cloud data backup
3. Information security measures
4. Database storage and management measures
5. Intellectual property rights in producing health education multimedia to protect medical staff
6. Functional interface of this automated intelligent education software system

Research steps The subjects are randomly assigned to the intervention group (receiving the automated intelligent education software system) and the control group (receiving the original medical care method), and the disease prognosis of the two groups is tracked six to twelve months after discharge (re- hospitalizations and deaths).

The following is a description of the admission and care process for the intervention group and the control groups:

1. Intervention group (accepting the operation process of automated intelligent education software system):

1. Execute registration and qualification review
2. Automated smart education interaction At the same time, the patient will receive a personal disease self-care education manual, and will get the contact number of the case manager in case the patients encounter emergencies or disease care needs at home (the patient can call for consultation on home care for diseases if the patient want).

2. Control group: After confirming that the diagnosis of heart failure is met, the patient will receive 10-15 minutes of disease care education from a nurse when the patient receives the case. At the same time, the patient will receive a personal disease self-care education manual, and will get the contact number of the case manager in case the patients encounter emergencies or disease care needs at home (the patient can call for consultation on home care for diseases if the patient want).

Data analysis Data are collected at 5 time points starting from enroll to 6 months. For assessment, a few questionnaires are used, including Heart Failure knowledge scale, self-care of heart failure index, hospital anxiety and depression scale, self-efficacy scale, quality of life scale and satisfaction scale. Data analysis is performed with SPSS 22.0 software. Statistical analysis includes descriptive statistics, cluster analysis, independent samples t-test, single factor Analysis of variance one-way ANOVA, and generalized estimating equations (generalized estimating equations, GEE).

ELIGIBILITY:
Inclusion Criteria：

* Patients with a diagnosis of heart failure
* Patients with age >= 20 years old
* patients with clear consciousness
* Patients who can communicate with by Chinese or Taiwanese, and are willing to participate this study

Exclusion Criteria：

* patients who are long-term bedridden, or living dependent of others
* patients who have severe psychological disease, or severe cognitive dysfunction
* patients without utilizing smartphone or internet

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite events of one-year Re-Hospitalization and all-cause death | 1 year
  Follow-up begins after enroll. Follow-up data are prospectively obtained every month from hospital records, personal communication with patients' physicians, telephone interviews, and records of regular visits to staff physicians' outpatient clinics. All-cause death is chosen as an endpoint because of the inter- relationship of heart failure with many other comorbidities in the patient cohort. Re-hospitalization is defined as a re-hospitalization due to worsening heart failure. In the statistical analysis for outcomes, composite events combining heart failure-related re-hospitalization and all-cause death will be estimated. Based on these two different endpoints, time to the first event was analyzed.
Heart Failure knowledge scale | 6 month
  The HF knowledge scale has 15 questions, self-administered questionnaire that covers items concerning HF knowledge in general, knowledge on HF treatment (including diet and fluid restriction) and HF symptoms and symptom recognition. For each item, patients can choose from three options, with one of the options being the correct answer. The scale has a minimum score of 0 (no knowledge) and a maximum score of 15 points (optimal knowledge).
Self-Care of Heart Failure Index (SCHFI) | 6 month
  SCHFI Version 6.2 has 22 items rated on a 4-point response scale, and divided into the following three scales: self-care maintenance, self-care management, and self-care confidence. The total score for each separate scale is standardized from zero to 100. Higher scores indicating higher contribution to self-care.
Hospital anxiety and depression scale (HADS) | 6 month
  The hospital anxiety and depression scale has 14 items. Seven of the items indicate anxiety and the remaining seven items indicate depression. The answer format offers four response options, which are scored with values ranging from 0 to 3. This results in scale values between 0 and 21 for each scale. The original test authors defined three ranges for both of the scales: 0-7 (non-cases), 8-10 (doubtful cases), and 11-21(cases).
Cardiac Self efficacy questionnaire | 6 month
  The core self-evaluations scale has 13 questions. A 5-point Likert scale was used, ranging from 1 (not at all confident) to 5 (very confident), a higher score indicates higher cardiac self-efficacy. Each question asks the patient to rate their level of confidence that using a five-point Likert scale. A score of 1 indicates "not at all", 2 "somewhat confident", 3 "moderately confident", 4 "very confident", and 5 "completely confident". The cardiac self-efficacy questionnaire has 13 items and the total score range is 0 to 65 points, with higher scores indicating greater self-efficacy.
Minnesota Living With Heart Failure questionnaire | 6 month
  The MLHF questionnaire is a disease-specific questionnaire designed to measure quality of life in patients with heart failure. This questionnaire is scored using a 5-point Likert scale and includes two subscales that address the physical and emotional domains, respectively. The questionnaire aims to reveal how patients feel about the changes in life caused by heart failure and symptom treatment during the past 1-month period. Each of the 21 questions in the questionnaire is scored from 0 to 5, with the total score range for the MLHF ranging from 0 to 105. Higher scores correlate with poorer quality of life.
Service satisfaction scale | 6 month
  The service satisfaction scale was developed by the researcher to understand the subjects' satisfaction with the use of the automated mobile education system or traditional outpatient care. It has 10 questions in total.

CONTACTS AND LOCATIONS:
Overall Officials: MIN-HUI LIU, RN, PhD, Principal Investigator — CHANG GUNG MEMORIAL HOSTIPAL, KEELUNG
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson L, Nordgren L. Heart Failure Patients' Perceptions of Received and Wanted Information: A Cross-Sectional Study. Clin Nurs Res. 2019 Mar;28(3):340-355. doi: 10.1177/1054773818787196. Epub 2018 Jul 10. PMID 29986617
- [Background] Arvanitaki A, Michou E, Kalogeropoulos A, Karvounis H, Giannakoulas G. Mildly symptomatic heart failure with reduced ejection fraction: diagnostic and therapeutic considerations. ESC Heart Fail. 2020 Aug;7(4):1477-1487. doi: 10.1002/ehf2.12701. Epub 2020 May 5. PMID 32368873
- [Background] Arestedt K, Saveman BI, Johansson P, Blomqvist K. Social support and its association with health-related quality of life among older patients with chronic heart failure. Eur J Cardiovasc Nurs. 2013 Feb;12(1):69-77. doi: 10.1177/1474515111432997. Epub 2012 Mar 28. PMID 22457369
- [Background] Austin RC, Schoonhoven L, Koutra V, Richardson A, Kalra PR, May CR. SYMptoms in chronic heart failure imPACT on burden of treatment (SYMPACT): a cross-sectional survey. ESC Heart Fail. 2022 Aug;9(4):2279-2290. doi: 10.1002/ehf2.13904. Epub 2022 Apr 21. PMID 35451208
- [Background] Allida S, Du H, Xu X, Prichard R, Chang S, Hickman LD, Davidson PM, Inglis SC. mHealth education interventions in heart failure. Cochrane Database Syst Rev. 2020 Jul 2;7(7):CD011845. doi: 10.1002/14651858.CD011845.pub2. PMID 32613635
- [Background] Bozkurt B, Coats AJ, Tsutsui H, Abdelhamid M, Adamopoulos S, Albert N, Anker SD, Atherton J, Bohm M, Butler J, Drazner MH, Felker GM, Filippatos G, Fonarow GC, Fiuzat M, Gomez-Mesa JE, Heidenreich P, Imamura T, Januzzi J, Jankowska EA, Khazanie P, Kinugawa K, Lam CSP, Matsue Y, Metra M, Ohtani T, Francesco Piepoli M, Ponikowski P, Rosano GMC, Sakata Y, SeferoviC P, Starling RC, Teerlink JR, Vardeny O, Yamamoto K, Yancy C, Zhang J, Zieroth S. Universal Definition and Classification of Heart Failure: A Report of the Heart Failure Society of America, Heart Failure Association of the European Society of Cardiology, Japanese Heart Failure Society and Writing Committee of the Universal Definition of Heart Failure. J Card Fail. 2021 Apr;27(4):387-413. doi: 10.1016/j.cardfail.2021.01.022. Epub 2021 Mar 1. PMID 33663906
- [Background] Checa C, Medina-Perucha L, Munoz MA, Verdu-Rotellar JM, Berenguera A. Living with advanced heart failure: A qualitative study. PLoS One. 2020 Dec 14;15(12):e0243974. doi: 10.1371/journal.pone.0243974. eCollection 2020. PMID 33315935
- [Background] Deek H, Newton PJ, Kabbani S, Hassouna B, Macdonald PS, Davidson PM. The Lebanese Heart Failure Snapshot: A National Presentation of Acute Heart Failure Admissions. J Nurs Scholarsh. 2020 Sep;52(5):506-514. doi: 10.1111/jnu.12583. Epub 2020 Aug 2. PMID 32741095
- [Background] Farwati M, Riaz H, Tang WHW. Digital Health Applications in Heart Failure: a Critical Appraisal of Literature. Curr Treat Options Cardiovasc Med. 2021;23(2):12. doi: 10.1007/s11936-020-00885-z. Epub 2021 Jan 16. PMID 33488049
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 May 3;79(17):e263-e421. doi: 10.1016/j.jacc.2021.12.012. Epub 2022 Apr 1. PMID 35379503
- [Background] Hearn J, Pham Q, Schwartz JI, Ssinabulya I, Akiteng AR, Ross HJ, Cafazzo JA. Lived Experiences and Technological Literacy of Heart Failure Patients and Clinicians at a Cardiac Care Centre in Uganda. Ann Glob Health. 2020 Jul 28;86(1):85. doi: 10.5334/aogh.2905. PMID 32832383
- [Background] Hiriscau EI, Bodolea C. The Role of Depression and Anxiety in Frail Patients with Heart Failure. Diseases. 2019 Jun 19;7(2):45. doi: 10.3390/diseases7020045. PMID 31248108
- [Background] Ivynian SE, Newton PJ, DiGiacomo M. Patient preferences for heart failure education and perceptions of patient-provider communication. Scand J Caring Sci. 2020 Dec;34(4):1094-1101. doi: 10.1111/scs.12820. Epub 2020 Jan 27. PMID 31985863
- [Background] Jones NR, Roalfe AK, Adoki I, Hobbs FDR, Taylor CJ. Survival of patients with chronic heart failure in the community: a systematic review and meta-analysis. Eur J Heart Fail. 2019 Nov;21(11):1306-1325. doi: 10.1002/ejhf.1594. Epub 2019 Sep 16. PMID 31523902
- [Background] Jeminiwa R, Hohmann L, Qian J, Garza K, Hansen R, Fox BI. Impact of eHealth on medication adherence among patients with asthma: A systematic review and meta-analysis. Respir Med. 2019 Mar;149:59-68. doi: 10.1016/j.rmed.2019.02.011. Epub 2019 Feb 15. PMID 30803887
- [Background] Kolasa J, Fraczek-Jucha M, Grabowski M, Jankowska EA, Lelonek M, Pawlak A, Uchmanowicz I, Nessler J. A quasi-experimental study examining a nurse-led educational program to improve disease knowledge and self-care for patients with acute decompensated heart failure with reduced ejection fraction. Adv Clin Exp Med. 2022 Mar;31(3):267-275. doi: 10.17219/acem/143989. PMID 34856078
- [Background] Kessing D, Denollet J, Widdershoven J, Kupper N. Psychological Determinants of Heart Failure Self-Care: Systematic Review and Meta-Analysis. Psychosom Med. 2016 May;78(4):412-31. doi: 10.1097/PSY.0000000000000270. PMID 27082055
- [Background] Lee KS, Cho YM, Oh SH, Jung MS, Yoon JY. Evaluation of the Heart Failure in Internet Patient Information: Descriptive Survey Study. Int J Environ Res Public Health. 2021 Jan 25;18(3):1047. doi: 10.3390/ijerph18031047. PMID 33503950
- [Background] Latifi M, Anvari Tafti M, Davari Dolatabadi N, Rafiei Z, Allahbakhshian Farsani L. E-Health: The Impact of Social Network on Self Care Behavior in Heart Failure Patients toward COVID-19 Epidemic. Adv Biomed Res. 2021 Jun 28;10:15. doi: 10.4103/abr.abr_195_20. eCollection 2021. PMID 34476223
- [Background] Lawrance L, McLeroy KR. Self-efficacy and health education. J Sch Health. 1986 Oct;56(8):317-21. doi: 10.1111/j.1746-1561.1986.tb05761.x. PMID 3534459
- [Background] Morken IM, Storm M, Soreide JA, Urstad KH, Karlsen B, Husebo AML. Posthospitalization Follow-Up of Patients With Heart Failure Using eHealth Solutions: Restricted Systematic Review. J Med Internet Res. 2022 Feb 15;24(2):e32946. doi: 10.2196/32946. PMID 35166680
- [Background] Rezakhani Moghaddam H, Ranjbaran S, Babazadeh T. The role of e-health literacy and some cognitive factors in adopting protective behaviors of COVID-19 in Khalkhal residents. Front Public Health. 2022 Jul 22;10:916362. doi: 10.3389/fpubh.2022.916362. eCollection 2022. PMID 35942262
- [Background] Graven LJ, Martorella G, Gordon G, Grant Keltner JS, Higgins MK. Predictors of depression in outpatients with heart failure: An observational study. Int J Nurs Stud. 2017 Apr;69:57-65. doi: 10.1016/j.ijnurstu.2017.01.014. Epub 2017 Feb 1. PMID 28182959
- [Background] Peyman N, Shahedi F, Abdollahi M, Doosti H, Zadehahmad Z. Impact of Self-Efficacy Strategies Education on Self-Care Behaviors among Heart Failure Patients. J Tehran Heart Cent. 2020 Jan;15(1):6-11. PMID 32742286
- [Background] Polikandrioti M, Kalafatakis F, Koutelekos I, Kokoularis D. Fatigue in heart failure outpatients: levels, associated factors, and the impact on quality of life. Arch Med Sci Atheroscler Dis. 2019 May 28;4:e103-e112. doi: 10.5114/amsad.2019.85406. eCollection 2019. PMID 31211277
- [Background] Petruzzo A, Paturzo M, Naletto M, Cohen MZ, Alvaro R, Vellone E. The lived experience of caregivers of persons with heart failure: A phenomenological study. Eur J Cardiovasc Nurs. 2017 Oct;16(7):638-645. doi: 10.1177/1474515117707666. Epub 2017 Apr 27. PMID 28447879
- [Background] Rector TS, Kubo SH, Cohn JN. Validity of the Minnesota Living with Heart Failure questionnaire as a measure of therapeutic response to enalapril or placebo. Am J Cardiol. 1993 May 1;71(12):1106-7. doi: 10.1016/0002-9149(93)90582-w. No abstract available. PMID 8475878
- [Background] Halbreich U. Theory and practice. Biol Psychiatry. 1990 Oct 15;28(8):649. doi: 10.1016/0006-3223(90)90450-g. No abstract available. PMID 1978688
- [Background] Scantlebury A, Booth A, Hanley B. Experiences, practices and barriers to accessing health information: A qualitative study. Int J Med Inform. 2017 Jul;103:103-108. doi: 10.1016/j.ijmedinf.2017.04.018. Epub 2017 May 1. PMID 28550995
- [Background] Sethares KA, Chin E, Jurgens CY. Predictors of delay in heart failure patients and consequences for outcomes. Curr Heart Fail Rep. 2015 Feb;12(1):94-105. doi: 10.1007/s11897-014-0241-5. PMID 25447709
- [Background] Shoemaker SJ, Wolf MS, Brach C. Development of the Patient Education Materials Assessment Tool (PEMAT): a new measure of understandability and actionability for print and audiovisual patient information. Patient Educ Couns. 2014 Sep;96(3):395-403. doi: 10.1016/j.pec.2014.05.027. Epub 2014 Jun 12. PMID 24973195
- [Background] Teng TK, Tromp J, Tay WT, Anand I, Ouwerkerk W, Chopra V, Wander GS, Yap JJ, MacDonald MR, Xu CF, Chia YM, Shimizu W; ASIAN-HF investigators; Richards AM, Voors A, Lam CS. Prescribing patterns of evidence-based heart failure pharmacotherapy and outcomes in the ASIAN-HF registry: a cohort study. Lancet Glob Health. 2018 Sep;6(9):e1008-e1018. doi: 10.1016/S2214-109X(18)30306-1. PMID 30103979
- [Background] Treskes RW, Van der Velde ET, Schoones JW, Schalij MJ. Implementation of smart technology to improve medication adherence in patients with cardiovascular disease: is it effective? Expert Rev Med Devices. 2018 Feb;15(2):119-126. doi: 10.1080/17434440.2018.1421456. Epub 2018 Jan 2. PMID 29271661
- [Background] Takeda A, Martin N, Taylor RS, Taylor SJ. Disease management interventions for heart failure. Cochrane Database Syst Rev. 2019 Jan 8;1(1):CD002752. doi: 10.1002/14651858.CD002752.pub4. PMID 30620776
- [Background] Sullivan MD, LaCroix AZ, Russo J, Katon WJ. Self-efficacy and self-reported functional status in coronary heart disease: a six-month prospective study. Psychosom Med. 1998 Jul-Aug;60(4):473-8. doi: 10.1097/00006842-199807000-00014. PMID 9710293
- [Background] van der Wal MH, Jaarsma T, Moser DK, van Veldhuisen DJ. Development and testing of the Dutch Heart Failure Knowledge Scale. Eur J Cardiovasc Nurs. 2005 Dec;4(4):273-7. doi: 10.1016/j.ejcnurse.2005.07.003. Epub 2005 Aug 29. PMID 16126459
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Zikmund V. Health--mental health--quality of life. Bratisl Lek Listy. 2001;102(11):527-9. PMID 11901711